CLINICAL TRIAL: NCT01137773
Title: Does Maintenance of Normoglycemia Change Neurological Outcome in Patients Recovering From Traumatic Brain Injury and Subarachnoid or Intraparenchymal Hemorrhage?
Brief Title: Normoglycemia and Neurological Outcome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rainer Lenhardt, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UofL IRB #562.06
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Acute, Non-traumatic Subarachnoid Hemorrhage; Intraparenchymal Hemorrhage; Brain Injuries
Keywords: SAH (Subarachnoid Hemorrhage); Brain Hemorrhage; Traumatic Brain Injury; SAH; ICH
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Intracranial Hemorrhages; Brain Injuries, Traumatic | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive IV Insulin (Experimental): Patients will receive IV insulin to maintain target glucose levels of 80-110 mg/dl
  Interventions: Drug: Insulin
- Conventional Insulin Treatment (Active Comparator): Patents will receive conventional IV insulin treatment with target glucose levels of 150-170 mg/dl
  Interventions: Drug: Conventional insulin treatment

INTERVENTIONS:
Drug: Insulin — All patients in the trial will have blood taken hourly for glucose analysis, regardless of their designated group. Adjustments of the insulin dose will be based on measurements of capillary blood glucose level.
  Arms: Intensive IV Insulin
Drug: Conventional insulin treatment — All patients in the trial will have blood taken hourly for glucose analysis , regardless of their designated group. Adjustments of the insulin dose will be based on measurements of capillary blood glucose level.
  Arms: Conventional Insulin Treatment

SUMMARY:
Brain injury patients who meet defined criteria will be assigned to intensive insulin treatment (target blood glucose levels of 10-110 mg/dl) or conventional IV insulin treatment (target glucose of 150-170 mg/dl). Follow up will occur at 3, 6 and 12 months. The primary outcome measure will be neurological outcome at 12 months according to Karnofsky Performance Scale (KPS). A general view of outcome will also be presented as favorable (good recovery+ moderate disability), unfavorable (severely disabled+ vegetative state), and dead.

Secondary outcome measures will be blood glucose levels and death.The investigators will also record systemic complications like pulmonary emboli, pulmonary edema, myocardial infarction, ventricular arrhythmias, and pneumonia.

DETAILED DESCRIPTION:
Demographic data, social and medical histories, and clinical features at onset will be obtained via patient or family interview shortly after admission . We want to get the patients enrolled in our protocol as soon as possible because we believe that hyperglycemia levels greater than 200 mg/dl is a secondary insult that should be prevented as early as possible. However, a twelve-hour period after ICU admission is necessary for initial diagnosis and assessment of the patient's status in order to identify the patient as a potential study subject and to get consent from the patient's legal representative.

Within twelve hours of ICU admission, qualifying patients will be randomized one of the two groups. Randomization will be based on computer-generated codes that will be maintained in sequentially numbered opaque envelopes. The randomization will be stratified according to the severity of neurological injury based on GCS. The three stratification groups will be GCS=6-8, GCS=9-11 and GCS=12-14. Randomization will be done using random sized blocks within stratum, and patients will be randomized within stratum to either:

1. Intensive intravenous insulin treatment (Target glucose levels of 80-110 mg/dl)
2. Conventional intravenous insulin treatment (Target glucose levels of 150-170 mg/dl)

All patients in the trial will have blood taken hourly for glucose analysis, regardless of their designated group. Adjustments of the insulin dose will be based on measurements of capillary blood glucose level. The interval between the glucose samples will be increased when patients satisfy discharge criteria from the intensive care unit. The insulin dose adjustments will be made by a team of intensive care nurses, assisted by a study nurse who is not otherwise involved in the clinical care of the patients. RBC transfusions, if necessary, will be administered one unit at a time, and the patient's hemoglobin concentration will be measured before and after each transfusion.

All patients enrolled in the study will receive saline infusion supplemented with potassium. An orogastric or nasogastric feeding tube (Dobhoff tube) will be inserted. Enteral feeding will be started per feeding protocol with the goal of starting on day one. After insertion of a nasogastric or orogastric tube, tube position will be verified with abdominal x-ray. Enteral feeding will be instituted with 25 to 30 nonprotein kilocalories per kilogram of body weight per 24 hours and a balanced composition (including 0.13 to 0.26 g of nitrogen per kilogram per 24 hours and 20 to 40 percent of nonprotein in the form of lipids). 69 Formula used will be recorded. Patients will be fed continuously starting at a rate of 25 ml/hour. If continuous enteral feeding cannot be instituted or has to be stopped and enteral nutrition is anticipated to be interrupted for more than 7 days, total parenteral nutrition will be initiated. Patients will be allowed to progress to a regular oral diet after they have passed a swallowing study.

The underlying neurological conditions will be managed by the neurosurgical team according to the protocols of the Department of Neurosurgery of the University of Louisville.

When participating patients' physiological statuses have stabilized and the need for ICU monitoring and care is no longer necessary, they will be discharged to a lower level of care (in accordance with the 1999 guidelines of Task Force of the American College of Critical Care Medicine, Society of Critical Care Medicine). Upon discharge from ICU, patients in all groups will be treated with subcutaneous insulin according to established transition guidelines.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic SAH, ICH, or TBI
* Glasgow Coma Scale between 6 and 14
* admitted to an ICU of University of Louisville Hospital

Exclusion Criteria:

* Patients <18 and >80 years
* GCS Motor score <4 or an overall GCS score of 15
* diabetic patients who suffer from dialysis-dependent diabetic nephropathy
* patients with multiple injuries
* patients who would have been classified as ASA 3 status prior to their acute neurological event

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive IV Insulin: Patients received target glucose levels of 80-110 mg/dl
- Conventional Insulin Treatment: Subjects received conventional (150-170 mg/dl) glucose control
Period: Overall Study
Arm/Group | Intensive IV Insulin | Conventional Insulin Treatment
Started | 33 | 23
Completed | 24 | 20
Not Completed | 9 | 3
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensive IV Insulin: Patients will received IV insulin to maintain target glucose levels of 80-110 mg/dl
- Convention Insulin Treatment: conventional (150-170 mg/dl, n = 20) glucose control
- Total: Total of all reporting groups
Arm/Group | Intensive IV Insulin | Convention Insulin Treatment | Total
Number analyzed (Participants) | 33 | 23 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 23 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 23 | 56

OUTCOME MEASURES:

1. Primary Outcome: Karnovsky Performance Status Scale of Functional Impairment
Description: The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. It can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. Patients are assigned a value from 0 to 100 based on the following definitions: Normal no complaints; no evidence of disease - 100. Normal activity with effort; some signs or symptoms of disease - 80. Requires occasional assistance, but is able to care for most of his personal needs - 60. Disabled; requires special care and assistance - 40. Very sick; hospital admission necessary; active supportive treatment necessary- 20. Dead- 0
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intensive IV Insulin | Convention Insulin Treatment
Number analyzed (Participants) | 24 | 20
units on a scale | 53 (55) | 60 (25)
Statistical Analysis 1: Comparison: Intensive IV Insulin vs Convention Insulin Treatment; Test type: Superiority; p = 0.49, t-test, 2 sided

2. Secondary Outcome: Blood Glucose Concentration
Description: average blood glucose concentration while the patients received insulin drip
Time Frame: 24 h
Measure: Mean (Standard Deviation); unit: mg/dl blood
Arm/Group | Intensive IV Insulin | Conventional Insulin Treatment
Number analyzed (Participants) | 24 | 20
mg/dl blood | 99 (9) | 138 (20)
Statistical Analysis 1: Comparison: Intensive IV Insulin; Test type: Superiority; p = .70, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Convention Insulin Treatment: target glucose levels of 150-170 mg/dl
Arm/Group | Intensive IV Insulin | Convention Insulin Treatment
All-Cause Mortality (participants affected / at risk) | 3/33 | 3/23
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/23
Other Adverse Events (participants affected / at risk) | 0/33 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes